CLINICAL TRIAL: NCT02981667
Title: Enjoyment Responses to High Intensity Interval Training and Moderate Intensity Continuous Exercise
Brief Title: Higher Enjoyment in Response to High Intensity Interval Training Versus Moderate Intensity Continuous Exercise
Status: Completed | Type: Observational
Sponsor: California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Todd A. Astorino Ph.D, Professor, Dept. of Kinesiology, California State University, San Marcos
Other Study IDs: astorino1
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Exercise Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active men and women: Healthy, active men and women ages 18-45 yr completed 1 bout of high intensity interval training and moderate intensity continuous training in a randomized, crossover design.
  Interventions: Other: Exercise intensity

INTERVENTIONS:
Other: Exercise intensity — Participants were randomized to 1 or 2 exercise intensities, moderate or high (interval training).

SUMMARY:
Previous research is equivocal concerning if high intensity interval training is viewed as more aversive versus moderate exercise. Our data in active men and women showed that interval training is viewed as more enjoyable than higher volume moderate exercise.

DETAILED DESCRIPTION:
Twelve men and women who were habitually active initially performed ramp exercise on a cycle ergometer to assess maximal oxygen uptake (VO2max) and peak power output (PPO), which was used to determine workload for the subsequent 2 bouts. They returned at least 48 h later at the same time of day to complete high intensity interval training (HIIT consisting of repeated 1 min bouts at 85 %PPO) or moderate intensity continuous training (MICT consisting of 25 min at 40 %PPO). During exercise, heart rate, oxygen uptake, perceived exertion, pleasure:displeasure, and blood lactate concentration were continuously assessed. Ten minutes post-exercise, physical activity enjoyment was measured. Data showed that despite higher oxygen uptake, heart rate, blood lactate concentration, and perceived exertion in HIIT, enjoyment was higher in HIIT versus MICT.

ELIGIBILITY:
Inclusion Criteria:

* Habitually active, healthy, non-obese

Exclusion Criteria:

* Sedentary, unhealthy, joint pain precluding tolerance to exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Habitually active young men and women ages 18-45 yr
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Physical activity enjoyment score (PACES) | This was measured 10 min post-exercise in all participants during the 3 mo of data collection.
  This is an 18-item categorical survey used to assess participants' enjoyment of the bout of physical activity that was just completed
Oxygen uptake | Measured continuously during exercise during the 3 mo of data collection.
  Oxygen uptake (VO2) represents mitochondrial consumption of oxygen to drive cellular metabolism generating ATP to support muscular contraction.

IPD SHARING:
Plan to Share IPD: No
Data are accepted for publication in PLoS One, an open-access journal, which makes the aggregate data available to all researchers.

REFERENCES:
- [Derived] Thum JS, Parsons G, Whittle T, Astorino TA. High-Intensity Interval Training Elicits Higher Enjoyment than Moderate Intensity Continuous Exercise. PLoS One. 2017 Jan 11;12(1):e0166299. doi: 10.1371/journal.pone.0166299. eCollection 2017. PMID 28076352